CLINICAL TRIAL: NCT06822907
Title: Immunogenicity and Safety of the 20-Valent Pneumococcal Conjugate Vaccine (PCV-20) Administered During an Acute Febrile Illness in Adults: a Multicentric Randomized Non-inferiority Trial
Brief Title: Immunogenicity and Safety PCV-20 of the Vaccine Administered During an Acute Febrile Illness in Adults
Acronym: PREV-HOSPIT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government); IREIVAC/COVIREIVAC Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19PH225; 2024-517411-73-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Febrile Illness; Pneumococcal Infections
Keywords: vaccin; pneumococcal; Prevenar 20; Acute febrile illness; infections; PCV-20; PCV-21
MeSH Terms: conditions — Pneumococcal Infections; Infections | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Prospective Randomised Open Blinded End-point trial (PROBE) Non inferiority design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early vaccination (Experimental): The patient will receive unique dose of the PCV-20 vaccine as soon as possible and until 72h after apyrexia.
  The "Prevenar 20" will be used
  Interventions: Biological: Early intervention
- Delayed vaccination (Active Comparator): From 15 days and until 58 days after fever resolution (i.e after the first day with a body temperature < 37.5°C without paracetamol use in the 6 previous hours) (whether or not the patient has been discharged) in the absence of fever, the patient will receive PCV-20 vaccination The "Prevenar 20" will be used
  Interventions: Biological: Delayed intervention

INTERVENTIONS:
Biological: Early intervention — In this arm, patient will receive unique dose of the PCV-20 vaccine (Prevnar 20) as soon as possible and until 72h after apyrexia.
  The "Prevenar 20" will be used Prevenar 20 will be injected by intramuscular route. The preferred site of injection is the deltoid muscle of the upper arm in adults.
  Arms: Early vaccination
Biological: Delayed intervention — In this arm, from 15 days and until 58 days after fever resolution (i.e after the first day with a body temperature < 37.5°C without paracetamol use in the 6 previous hours) (whether or not the patient has been discharged) in the absence of fever, the patient will receive unique dose of the PCV-20 vaccine (Prevnar 20).
  The "Prevenar 20" will be used Prevenar 20 will be injected by intramuscular route. The preferred site of injection is the deltoid muscle of the upper arm in adults.
  Arms: Delayed vaccination

SUMMARY:
Streptococcus pneumoniae is responsible for serious infections associated to numerous hospitalizations and high rate of mortality. The incidence and therefore the burden of pneumococcal infections have been significantly reduced thanks to the use of pneumococcal conjugate vaccines (PCVs). PCVs were shown to be effective against vaccine-type serotypes causing both non-invasive and invasive pneumococcal diseases (IPD) in children and adults. PCVs use in children was shown to have an impact on IPD incidence among adults due to herd immunity and on antimicrobial resistance. To increase the protection of at-risk patients against IPD, the 20-valent PCV (PCV-20) is recently recommended in adults, after a period where PCV-13 followed by pneumococcal polysaccharide vaccine 23 valent (PPV-23) was recommended. PCV-20 effectiveness against IPD and against pneumonia was inferred from immunobridging with PCV-13. Indeed PCV-13 was shown effective to reduce the incidence of low respiratory tract infections and IPD (bacteraemia and meningitis) in 65-years-old-adults and older. Currently immunization against S. pneumoniae is recommended with PCV-20 for adult patients at-risk for IPD such as immunocompromised (=high-risk patients) and in immunocompetent people with underlying chronic conditions (cardiovascular, liver, pulmonary, kidney diseases and diabetes mellitus) (=medium risk patients). However, vaccine coverage against IPD in adults remains low globally, and does not exceed 5 % in France. Reducing missed opportunities of vaccination for S. pneumoniae is crucial.

DETAILED DESCRIPTION:
Patients at-risk of IPD are very frequently hospitalized for acute febrile illnesses. More than 50 % of the IPD at-risk patients hospitalized for an IPD or a pneumonia have been admitted to the hospital during the past 5 years without receiving a pneumococcal vaccination. Hospitalization appears to be therefore an opportunity to provide vaccines. However, physicians usually consider that vaccines should be postponed during an acute febrile illness including if non-severe. This consideration of not vaccinating during an acute febrile illness is however not evidence-based. This is associated to concerns about a potential risk of an impaired response to the vaccine and safety. In children, data about vaccination during a febrile illness have shown no safety nor efficacy concerns. In most countries, recommendations regarding this particular point are unclear.

In fine, vaccination is then rarely provided during the hospital stay as well as after discharge including in the USA, a country where it is recommended to vaccinate whatever the body temperature is and during hospitalization. Reluctance to immunize adults in this situation is probably due to the absence of evidence showing that it is as effective and safe as vaccinating patients without an acute or febrile illness.

To reduce the number of missed opportunities to immunize adults against S. pneumoniae, investigators aim to demonstrate that the administration of PCV-20 during an acute non-severe febrile illness is non-inferior than the administration one month after fever resolution in terms of immunogenicity (assessed by vaccine types (VT) Immunoglobulin G (IgG) concentrations and at least 2-fold change increase), and that it is as safe.

ELIGIBILITY:
Inclusion criteria :

* History of body temperature ≥ 38°C measured at least twice prior to randomization (Randomization must be performed as soon as possible on a febrile patient or 72 hours after apyrexia at the latest)
* Having at least one comorbidity that defines patients as medium or high risk for pneumococcal invasive infection:

  * Medium risk: Cyanogenic congenital heart disease; chronic heart failure; chronic respiratory failure; chronic obstructive pulmonary disease; emphysema; severe asthma under chronic treatment; chronic renal failure; chronic liver disease; diabetes mellitus treated; Osteo-meningeal leak or cochlear implant; Age > 65 years old.
  * High risk : Hypo or asplenic people; hereditary immunodeficiency syndromes; people living with HIV; solid organ transplanted; People under immunosuppressors (corticosteroids, biotherapy) for an auto-immune or an inflammatory chronic disease; patients with nephrotic syndrome
* Hospitalization for > 24 hours long
* Social security affiliation
* Signed informed consent

Exclusion criteria :

* Patient unable to give informed consent
* Curators, wardship
* History of previous vaccination with PCV-7 or PCV-13 or PCV-20
* History of PPV-23 in the previous year
* Patient having received another vaccination within one month prior to inclusion or planning another vaccination in the month after inclusion except for Influenza vaccine.
* Patient with history of bone marrow transplantation
* Patient with haematological malignancies
* Patient under chemotherapy for solid tumor or with a history of chemotherapy in the past three months
* Patient treated with Rituximab currently or in the past 6 months
* Patient with Sequential Organ Failure Assessment (qSOFA ) score ≥ 2 at randomization (acute severe febrile illness)
* Patient hospitalized in an Intensive Care Unit
* Pregnancy
* Breastfeeding woman
* Recipients of polyclonal gammaglobulins in the past three months
* Inability to follow the protocol
* Bleeding disorder contra-indicating intramuscular injection according to the investigator
* History of allergy to PCV-20 or vaccine-related components.
* S. pneumoniae infection with laboratory confirmation (blood culture, culture from a sterile site, urinary or Cerebrospinal fluid antigens, sputum culture with > 10^7 colony forming unit (CFU)/mL) being the cause of the current hospitalization

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of immune "good responders" to PCV-20 in both arms | 1 month post vaccination
  Good responders is defined as - a seroconversion (a 2-fold increase in VT IgG after vaccination), for ≥10 vaccine serotypes (VT) among the 13 tested on 20 in ELISA, AND an immune protective response defined as ELISA IgG > 1,3 μg/mL in ≥ 10 out 13 VT.
  OR
  - -a seroconversion (a 4-fold increase in VT IgG after vaccination), for ≥10 vaccine serotypes (VT) among the 13 tested on 20 in ELISA, AND an immune protective response defined as ELISA IgG < 1,3 μg/mL in ≥ 10 out 13 VT.

SECONDARY OUTCOMES:
Safety endpoints in both arms in the month following vaccination : adverse events | 1 month post vaccination
  Number, type and severity of solicited (in the 7 days following vaccination) and unsolicited (in the month following vaccination) adverse events
Frequency of local reactions | 1 month post vaccination
  Local reactions will be defined as : pain, redness, and swelling at the study vaccine injection site and limitation of arm movement
Frequency of systemic events related to the vaccination | 1 month post vaccination
  Onset or worsening of fever, diarrhoea, chills, fatigue, headache, vomiting, decreased appetite, rash, muscle pain, joint pain). An independent blinded central adjudication committee will define the onset or worsening of symptoms and will review all systemic events.
Proportion of immune good responders serotype by serotype | 1 month post vaccination
  "Good responders" being defined above (primary end-point)
  A blood sample for immunologic analysis will be performed
opsonophagocytic activity (OPA) IgG titers for serotype by serotype | 1 month post vaccination
  A blood sample for immunologic analysis will be performed. ELISA method will be used for immunologic analysis.
Proportion of the participants immune "good responders" to PCV-20 in both arms. | 1 year post vaccination
  "Good responders" being defined above (primary end-point) A blood sample for immunologic analysis will be performed. ELISA method will be used for immunologic analysis.
Number of low respiratory tract infections events | 1 year post vaccination
  Data about occurrence of respiratory infections will be recorded.
Number of confirmed S.pneumoniae infections | 1 year post vaccination
  Data about pneumococcal infection will be recorded.
Analyze the gut microbiota on the immune response | 1 year post vaccination
  Analyze the gut microbiota on the immune response in both arm ( during an acute febrile illness or 15-58 days after resolution of the acute febrile illness)
  A stool sample is taken before vaccination
Reactogenic inflammatory response after vaccination | 1 month post vaccination
  Fold change kinetics (transcriptomics) (before and at 24 hours after vaccination) of vaccine-induced gene signatures in peripheral blood mononuclear cells and serum cytokine levels at baseline and 24 hours after vaccination in both arms.
Frequency of specific PCV-20 interferon-gamma (IFNg) secreting CD4 or CD8 T cells | 1 month post vaccination
  Blood sample will be collected 1 month post-vaccination.
Frequency of specific PCV-20 IFNg secreting CD4 or CD8 T cells | 1 year post vaccination
  Blood sample will be collected 1 year post-vaccination.
Proportion of volunteers with circulatory immunoglobulin A (IgA) | 1 month post vaccination
  Blood sample will be collected 1 month post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth BOTELHO-NEVERS, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (24):
- France (24):
  - CHU de Saint-Etienne, Saint-Etienne, France
  - Centre Hospitalier, Annecy
  - Centre Hospitalier Universitaire, Besançon
  - Centre Hospitalier, Bordeaux
  - Centre Hospitalier Universitaire, Brest
  - Centre Hospitalier, Brest
  - Centre Hospitalier General Metropole Savoie, Chambéry
  - Centre Hospitalier de Creteil, Créteil
  - Centre Hospitalier Universitaire, Dijon
  - Centre Hospitalier Universitaire, Grenoble
  - Centre Hospitalier, La Roche-sur-Yon
  - Centre Hospitalier General, Le Mans
  - Centre Hospitalier, Le Puy-en-Velay
  - Centre Hospitalier Universitaire, Lille
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Regional Universitaire, Montpellier
  - Centre Hospitalier Universitaire, Nancy
  - Centre Hospitalier Universitaire, Nantes
  - Centre Hospitalier Universitaire, Nice
  - Centre Hospitalier Universitaire, Nîmes
  - Centre Hospitalier Bichat, Paris
  - Assistance Publique Hopitaux de Paris, Paris
  - Centre Hospitalier Universitaire, Rennes
  - Centre Hospitalier Universitaire, Rouen

IPD SHARING:
Plan to Share IPD: No